CLINICAL TRIAL: NCT03560895
Title: Ultrasonographic Prediction of Actual Tube Size and Performance Characteristics of Cuffed Vs Un-Cuffed Endotracheal Tubes in Pediatric Surgical Patients.
Brief Title: US Prediction of Actual Tube Size and Performance Characteristics of Pediatric Cuffed Vs Un-Cuffed ETT.
Acronym: USETT
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Professor of anesthesia and intensive care, faculty of medicine, Assiut university., Assiut University
Other Study IDs: 17200201
Record Dates: First submitted 2018-06-05; First posted 2018-06-18 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Airway Complication of Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group I: Patients will be anesthetized using high-volume low-pressure cuffed endotracheal tube (Flexicare-UK) ) with its outer diameter determined by ultrasonography.
  Interventions: Device: cuffed endotracheal tube
- Group II: Patients will be anesthetized using uncuffed endotracheal tube (Flexicare-UK) with its outer diameter determined by ultrasonography.
  Interventions: Device: Uncuffed endotracheal tube

INTERVENTIONS:
Device: cuffed endotracheal tube — Patients will be anesthetized using high-volume low-pressure cuffed endotracheal tube
  Other Names: C ETT
  Groups: Group I
Device: Uncuffed endotracheal tube — Patients will be anesthetized using uncuffed endotracheal tube
  Other Names: ETT
  Groups: Group II

SUMMARY:
The aim of this study will be to test the accuracy of Sonography in determining the endotracheal tube size in pediatric patients whether cuffed or un-cuffed.

DETAILED DESCRIPTION:
* Children's tracheas have traditionally been intubated with un-cuffed tracheal tubes (TT) due to differences between adult and pediatric sub-glottic anatomy and fears that cuffs may lead to mucosal damage and subglottic stenosis. Despite this, cuffed TTs are increasingly used in pediatric anesthesia. Over the last 20 years, evidence suggests that cuffed TT may have advantages over un-cuffed, and are associated with at least similar, if not superior, airway outcomes when compared with un-cuffed TT in children.
* Formulas based on age and height often fail to reliably predict the proper endotracheal tube (ETT) size in pediatric patients. Visualization of the pediatric subglottic airway diameter by ultrasonography (USG) can enable a practitioner to better predict ETT size, preventing unnecessary tube changes and airway trauma. Also, Visualization of the transvers diameter of epiphyseal end of distal radius by ultrasonography (USG) has been recently investigated and can enable a practitioner to better predict ETT size. Recent reports suggest that the diameter of the subglottic upper airway can be determined by ultrasonography in healthy young adults and pediatric patients . However, the extent to which ultrasonography by these two measurements can predict optimal ETT size in pediatric patients remains under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Weight: 10-30 kg.
* Age: 1-6 years.
* Sex: both males and females.
* ASA physical status: I-II.
* Operation: elective surgery in which airway management with an endotracheal tube is needed.

Exclusion Criteria:

* Upper airway malformations.
* Upper airway surgery.
* Active respiratory illness (cough, fever, rhinorrhea) on the day of anesthesia,
* Anticipated difficult airway.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1-6 years of both sexes undergoing surgical procedures in which an endotracheal tube is needed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
The rate of agreement between the reference tube size based on sonographic measurements and the final BEST-FIT ETT | AT induction of anesthesia
  The rate of agreement between the reference tube size based on sonographic measurements and the final BEST-FIT ETT

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdelghaffar, MD, Principal Investigator — Professor of anesthesia, faculty of medicine, Assiut university, Egypt.
Locations (1):
- Pediatric hospital, faculty of medicine, Assiut university, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No